CLINICAL TRIAL: NCT06383013
Title: Phase II Study to Evaluate the Efficacy and Safety of Topical BB-101 for the Treatment of Diabetic Lower Leg and Foot Ulcers
Brief Title: BB-101 for the Treatment of Diabetic Lower Leg and Foot Ulcers
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Blue Blood Biotech Corp. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BB-101-BBCBB1A
Record Dates: First submitted 2024-04-22; First posted 2024-04-25 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2024-08

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- High Dose Dosing Group (Active Comparator): High Dose BB-101 topical solution will be applied on the target lower leg or foot ulcer once a for for 4 consecutive weeks.
  Interventions: Biological: BB-101
- Low Dose Dosing Group (Active Comparator): Low Dose BB-101 topical solution will be applied on the target lower leg or foot ulcer once a for for 4 consecutive weeks.
  Interventions: Biological: BB-101
- Placebo Dosing Group (Placebo Comparator): Placebo will be applied on the target lower leg or foot ulcer once a for for 4 consecutive weeks.
  Interventions: Biological: BB-101

INTERVENTIONS:
Biological: BB-101 — Subjects will be randomized to receive BB-101 or placebo, and expected 32 subjects for each arm.

SUMMARY:
This is a randomized, double-blinded, vehicle-controlled, parallel, phase II study to evaluate the efficacy and safety of topical BB-101 for the treatment of diabetic lower leg and foot ulcer.

DETAILED DESCRIPTION:
This is a randomized, double-blinded, vehicle-controlled, parallel, phase II study to evaluate the efficacy and safety of topical BB-101 for the treatment of diabetic lower leg and foot ulcer.

All subjects will receive standard-of-care ulcer treatment from screening through the last study visit.

The study will be conducted at multiple investigational sites located in Taiwan. Additional sites and countries may be added during the course of the study if required.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, at least 20 years of age (inclusive) at the date of Screening
* Subject or legally authorized representative who is able to understand the nature of this study and accepts to enter the study by signing written informed consent
* Subject agrees to comply with ulcer care regimen for the duration of the study and is willing to return for all mandatory visits as defined in the protocol
* Subject with Type 1 or Type 2 diabetes mellitus (criteria for the diagnosis of diabetes mellitus per American Diabetes Association) and is under the care of a physician for the management of diabetes mellitus
* Subject with glycosylated hemoglobin (HbA1c) ≤ 12%
* Subject with at least one diabetic foot ulcer meets the following criteria at Screening

Visit:

i. Located below knees; ii. Not healing for ≥ 4 weeks prior to Screening Visit despite appropriate care; iii. Ulcer size of ≥ 1 cm2 to ≤ 10 cm2 measured by the electronic measuring device following sharp debridement (if necessary) at Screening Visit and reconfirmed at Randomization Visit; iv. The largest ulcer will be selected as target ulcer. If ≥ 2 ulcers have the largest size, the one with the worst grade by Wagner Classification will be selected. If ≥ 2 ulcers have the largest size and grade, the one with longest duration will be selected; v. The target ulcer is classified as Grade 1 to Grade 2 according to Wagner Classification System for diabetic foot ulcer; vi. The target ulcer should be without clinical signs and symptoms of infection

* Subject with adequate circulation to the affected lower limb, as demonstrated by at least one of the following criteria: i. Dorsum transcutaneous oximetry (TcPO2) ≥ 30 mmHg ii. Ankle brachial pressure index (ABPI) ≥ 0.7 iii. Absolute toe blood pressure > 30 mmHg iv. Doppler ultrasonography showed < 75% stenosis in the lower extremity arteries
* Subject with adequate hepatic and renal function:

  i. Serum creatinine ≤ 3 mg/dL ii. ALT and AST ≤ 2 × ULN
* Subject with adequate hematology function:

  i. Absolute neutrophil count (ANC) ≥ 1,500 cells/μL ii. Total white blood cell (WBC) ≥ 3,000 cells/μL iii. Platelets ≥ 100,000 counts/μL iv. Hemoglobin ≥ 10 g/dL for male, ≥ 9 g/dL for female
* Female subjects show negative serum pregnancy test results within 21 days prior to the first study treatment.
* All male subjects and female subjects with child-bearing potential (between puberty and 2 years after menopause) should use at least any one of the appropriate contraception methods during dosing and for at least 4 weeks after stopping study treatment.

Exclusion Criteria:

* Clinical signs and symptoms of infection of target ulcer assessed by clinical evaluation.

The presence of infection is defined by ≥ 2 of the items presented as:

* Local swelling or induration
* Erythema > 0.5 cm around wound
* Local tenderness or pain
* Local increased warmth
* Purulent discharge

  * Subject with cellulitis or gangrene on the lower leg or foot with the target ulcer
  * Subject with active osteomyelitis
  * With target ulcer size decreased or increased by at least 30% after receiving 2 weeks of standard-of-care for diabetic foot ulcer before Randomization visit
  * Subject with another open ulcer < 2 cm away from target ulcer, on the same lower leg or foot
  * Subject with target ulcer caused primarily by etiologies not related to diabetes
  * Subject with target ulcers related to an incompletely healed amputation wound
  * Subject with any structural deformity of the lower leg or foot under study that would prevent off-loading of the target ulcer; subject with conditions which may interfere the off-loading effect may be excluded by the Investigators' judgment
  * Subject is scheduled to (or has received within 4 weeks prior to Screen Visit) receive any of the following medications or treatments:
* Platelet-derived product (e.g., becaplermin) or other growth factors on the target ulcer
* Systemic corticosteroids (other than for inhalation), immunosuppressive agents, radiation therapy, or chemotherapeutic agents
* Participation in a clinical trial of an investigational drug or device

  * Previous use of autologous graft or allogeneic graft, or dermal substitute or living skin equivalent (e.g., Dermagraft® or Apligraf® ) on the target ulcer or hyperbaric oxygen therapy within 2 weeks prior to Screening Visit
  * Use of any topical antimicrobials or enzymatic debridement treatment to treat the target ulcer within 7 days prior to Screening Visit
  * Subject with history of cancer or current cancer, with the exception of basal cell carcinoma, squamous cell carcinoma in situ of the skin, or cervical carcinoma in situ that has been treated with no evidence of recurrence, or squamous cell carcinoma of the skin that has been treated with no evidence of recurrence within 5 years prior to administration of any study agent
  * Vasculitis, connective tissue diseases, or any medical conditions known to impair ulcer healing, other than diabetes
  * Subject diagnosed with sickle cell disease
  * Subject with clinically significant electrocardiogram (ECG) abnormality, as determined by the Investigator
  * Poor nutritional status (serum albumin < 2.5 g/dL)
  * C-reactive protein (CRP) > 50 mg/dL
  * Subject had a history of drug abuse or alcohol abuse according to the Diagnostic and Statistical Manual of Mental Disorders 5th edition (DSM-5) criteria.
  * Patient with positive result of Human immunodeficiency virus (HIV)
  * Female subject in lactation during the study period
  * Subject with underlying medical, mental or psychological conditions that would impair the treatment compliance, or in the opinion of the Investigator would not permit to participate in the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy Evaluation | 4 weeks
  Percent change in wound surface area (cm^2) at each visit from baseline

SECONDARY OUTCOMES:
Safety Evaluation | 6 weeks
  To evaluate the Laboratory data, ECG examination results, physical examinations and vital signs changes from baseline, and AE incidences
Secondary Efficacy Evaluation | 4 weeks
  Incidence of complete wound closure and change in Wagner Scale

OTHER OUTCOMES:
Exploratory Objectives | 6 weeks
  Percent surface area of wound covered by granulation tissue
Exploratory Objectives | 6 weeks
  Change of ulcer conditions

CONTACTS AND LOCATIONS:
Overall Officials: Shug-Cheng Chang, MD, Principal Investigator — Taipei Medical University-Shuang Ho Hospital,Ministry of Health and Welfare
Locations (1):
- Taipei Medical University-Shuang Ho Hospital,Ministry of Health and Welfare, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No